CLINICAL TRIAL: NCT06720714
Title: An Open-Label, Single-Dose Study to Assess the Concentration of Rozanolixizumab in the Breast Milk of Healthy Lactating Women
Brief Title: A Study to Assess the Concentration of Rozanolixizumab in the Breast Milk of Healthy Lactating Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP0141
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Healthy Participants
Keywords: Phase 1; Healthy lactating women; rozanolixizumab; UCB7665
MeSH Terms: interventions — rozanolixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rozanolixizumab arm (Experimental): Study participants enrolled in this arm will receive a single dose of subcutaneous rozanolixizumab
  Interventions: Drug: Rozanolixizumab

INTERVENTIONS:
Drug: Rozanolixizumab — Dose formulation: Solution for injection Route of administration: Subcutaneous infusion
  Other Names: UCB7665

SUMMARY:
The purpose of the study is to assess the concentration of rozanolixizumab in mature breast milk of healthy study participants following administration of a single dose of rozanolixizumab

ELIGIBILITY:
Inclusion criteria

* Study participant must be minimum 18 years at the time of signing the informed consent form (ICF)
* Study participant is lactating and will be at least 6 weeks postpartum on Day 1 of the study
* Study participant has voluntarily decided, prior to having knowledge of this study, to cease breast milk feeding (by any means) in relation to her current period of lactation. Study participant agrees to cease or suspend breast milk feeding by Day 1 of the study and to not resume breast milk feeding (by any means) or donate expressed breast milk for 8 weeks following administration of rozanolixizumab. Participants may decide to resume breast milk feeding 8 weeks after administration of rozanolixizumab, with the agreement that any breast milk collected (to maintain milk supply) during that 8-week period will be discarded
* Study participant is female

A female participant is eligible to participate if she is not pregnant and at least 1 of the following conditions applies:

* A woman of childbearing potential (WOCBP) who agrees to follow the contraceptive guidance during the Sampling Period and for at least 1 week after the last dose of study treatment OR
* Not a WOCBP (ie, premenopausal female with documented hysterectomy, documented bilateral salpingectomy, or documented bilateral oophorectomy)

Exclusion criteria

* Study participant has history of breast implants, breast augmentation, or breast reduction surgery
* Study participant has received live vaccine(s) within 4 weeks prior to Screening or plans to receive such vaccines during the study
* Study participant has received treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Study participant has had exposure to more than 3 new chemical entities within 12 months prior to dosing
* Study participant has had an active clinically significant infection within the last 6 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will enroll adult (≥18 years of age) healthy lactating women.
Enrollment: 15 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Concentration of rozanolixizumab in breast milk over a 7-day Sampling Period | From Day 1, 2, 3, 4, 5, 6 Visit up to Day 7 Visit.
  The breast milk collection and sampling time points will be: within 30 minutes predose and at 0 to ≤3, ≤6, ≤9, ≤12, ≤24, ≤36, ≤48, ≤60, ≤72, ≤84, ≤96, ≤108, ≤120, ≤132 and ≤144 hours (Day 7) after the start of infusion.

SECONDARY OUTCOMES:
Estimated daily infant dosage | From Day 1, 2, 3, 4, 5, 6 Visit up to Day 7 Visit.
  The estimated daily infant dosage of rozanolixizumab from breast milk will be calculated based on the concentration of rozanolixizumab in mature human breast milk for the Pharmacokinetic Set (PKS).
Relative infant dose of rozanolixizumab from breast milk | From Day 1, 2, 3, 4, 5, 6 Visit up to Day 7 Visit.
  The relative infant dose of rozanolixizumab from breast milk will be calculated as: Estimated daily infant dosage (mg/kg/day)/maternal dosage (mg/kg/day) x 100%
Occurrence of TEAEs | From Day 1 Visit up to the Safety Follow-Up Visit (Week 9)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Treatment emergent adverse events (TEAEs) are adverse events not present prior to the pharamceutical product administration or an already present event that worsens either in intensity or frequency

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (2):
- United States (2):
  - UP0141 2, San Antonio, Texas
  - UP0141 1, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, individual participant-level data cannot be adequately anonymized as there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.